CLINICAL TRIAL: NCT03548701
Title: Thromboelastometry Prediction Utility for Risk of Abortion
Acronym: TEMPURA
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Patrick Maher, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 18-0104
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Pregnancy Trimester, First; Abortion, Threatened
Keywords: Thromboelastometry; Vaginal Bleeding; Early Pregnancy
MeSH Terms: conditions — Abortion, Threatened; Uterine Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood collected at time of subject enrollment for thromboelastometry testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergency Department: Patients enrolled in the Emergency Department undergoing evaluation for threatened abortion abnormalities.
  Interventions: Diagnostic Test: Thromboelastometry testing
- Obstetric Clinic: Patients with normal pregnancies being treated at first obstetric visit in clinic.
  Interventions: Diagnostic Test: Thromboelastometry testing

INTERVENTIONS:
Diagnostic Test: Thromboelastometry testing — Thromboelastometry testing - a form of testing in whole blood for coagulation abnormalities

SUMMARY:
This study will use thromboelastometry in ED patients with vaginal bleeding, as well as healthy pregnant controls, to determine if abnormal results are associated with the presence of vaginal bleeding as well as later complications during pregnancy.

DETAILED DESCRIPTION:
First, a case control study with samples collected from patients in the ED and OB clinic at Mount Sinai Hospital will be performed. Blood samples are being collected at time of study entry. Patient health history will be collected and blood samples will be tested using thromboelastometry in prospective fashion. Samples will be compared between groups.

A prospective cohort will then be established using the subjects from the case control study. The purpose of this prospective cohort will be to collect outcomes of pregnancies to determine association with the initial thromboelastometry results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include pregnant women seen in the ED and OB clinic.

The ED patients will include those seen for vaginal bleeding during pregnancy at less than 20 weeks gestation.

OB Clinic patients will include those seen for first prenatal visit at which blood draw is performed, as long as this is also within 20 weeks estimated gestational age.

Exclusion Criteria:

* Patients with known histories of recurrent miscarriage, previously diagnosed thrombophilia, or other coagulopathy will be excluded.
* Patients with ectopic pregnancies will also be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known histories of recurrent miscarriage, previously diagnosed thrombophilia, or other coagulopathy will be excluded. Patients with ectopic pregnancies will also be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Maximum Clotting Firmness (MCF) | Day 1
  Thromboelastometry measurement of the Maximum Clot Firmness over the duration of the test. Performed as part of InTEM (response to ellagic acid) and ExTEM (response to tissue factor) measures.

SECONDARY OUTCOMES:
Clot formation time (CFT) | Day 1
  Time to thromboelastometry measurement of the angle between formation of clot at 0mm and 20mm of strength. Performed as part of InTEM (response to ellagic acid) and ExTEM (response to tissue factor) measures.
Clotting Time (CT) | Day 1
  Thromboelastometry measurement of the time to first clot formation. Performed as part of InTEM (response to ellagic acid) and ExTEM (response to tissue factor) measures.
Pregnancy Outcome | Within 40 weeks of enrollment at completion of pregnancy
  Assessment of pregnancy outcome. Variable is treated as categorical and coded as spontaneous abortion, preterm labor, or term labor.
Number of Pregnancy Complications | Within 40 weeks of enrollment at completion of pregnancy
  Number of Pregnancy complications as a composite including pre-eclampsia, postpartum hemorrhage, or other clotting or bleeding dysfunction such as pulmonary embolus or preterm bleeding episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Maher, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

REFERENCES:
- [Background] Weiss JL, Malone FD, Vidaver J, Ball RH, Nyberg DA, Comstock CH, Hankins GD, Berkowitz RL, Gross SJ, Dugoff L, Timor-Tritsch IE, D'Alton ME; FASTER Consortium. Threatened abortion: A risk factor for poor pregnancy outcome, a population-based screening study. Am J Obstet Gynecol. 2004 Mar;190(3):745-50. doi: 10.1016/j.ajog.2003.09.023. PMID 15042008
- [Background] Harville EW, Wilcox AJ, Baird DD, Weinberg CR. Vaginal bleeding in very early pregnancy. Hum Reprod. 2003 Sep;18(9):1944-7. doi: 10.1093/humrep/deg379. PMID 12923154
- [Background] Rai R, Tuddenham E, Backos M, Jivraj S, El'Gaddal S, Choy S, Cork B, Regan L. Thromboelastography, whole-blood haemostasis and recurrent miscarriage. Hum Reprod. 2003 Dec;18(12):2540-3. doi: 10.1093/humrep/deg494. PMID 14645169
- [Background] Bennett SA, Bagot CN, Appiah A, Johns J, Ross J, Roberts LN, Patel RK, Arya R. Women with unexplained recurrent pregnancy loss do not have evidence of an underlying prothrombotic state: experience with calibrated automated thrombography and rotational thromboelastometry. Thromb Res. 2014 May;133(5):892-9. doi: 10.1016/j.thromres.2014.02.002. Epub 2014 Feb 11. PMID 24613698
- [Background] Armstrong S, Fernando R, Ashpole K, Simons R, Columb M. Assessment of coagulation in the obstetric population using ROTEM(R) thromboelastometry. Int J Obstet Anesth. 2011 Oct;20(4):293-8. doi: 10.1016/j.ijoa.2011.05.004. Epub 2011 Aug 10. PMID 21835606